CLINICAL TRIAL: NCT05678842
Title: Balance Parameters and Weight Distributions at Different Kneeling Positions
Brief Title: Balance and Weight Distributions at Kneeling
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ferhat Öztürk, Principal Investigator, Hacettepe University
Other Study IDs: GO 22/124
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Balanced; Weight, Body
Keywords: kneeling; weight distribution; balance; lower extremity; asymmetry
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Descriptive — Descriptive

SUMMARY:
This study aims to examine balance parameters and weight distributions at different kneeling positions.

DETAILED DESCRIPTION:
A cross-sectional study design was used to describe the balance parameters and weight-bearing distributions on knee in different kneeling positions with different ankle conditions. The participants signed informed consent forms before the study was performed on a voluntary basis. Inclusion criteria were defined as being between 18-30 years old and not having knee pain with kneeling. Exclusion criteria were previous history of lower limb pain/pathology, trauma, and/or surgery, any neurological, rheumatological or oncological disorders that would affect balance, have performed high intensity physical activities last 72 hours before test day, and BMI > 25. Balance parameters and weight distribution to each knee were evaluated three times at upright kneeling (UK) and full kneeling (FK) positions, in different ankle conditions (dorsiflexion and plantarflexion) with static balance device. Test-retest ICC values were calculated for all procedures.

ELIGIBILITY:
Inclusion Criteria:

* being between 18-30 years old
* not having knee pain with kneeling

Exclusion Criteria:

* previous history of lower limb pain/pathology,
* trauma, and/or surgery, any neurological, rheumatological or oncological disorders that would affect balance,
* have performed high intensity physical activities last 72 hours before test day,
* BMI > 25

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
To investigate balance parameters (postural sway (mm) ) in different kneeling positions. | one year
  Balance parameters and weight distribution to each knee were evaluated three times at upright kneeling (UK) and full kneeling (FK) positions, in different ankle conditions (dorsiflexion and plantarflexion) with static balance device. HurSmart balance system (HUR smart balance, HUR, Helsinki, Finland) was used for assessed the static balance. Postural sways to antero-posterior (A-P) and medio-lateral (M-L) directions were calculated.
weight distributions (kg) in different kneeling positions. | one year
  weight distribution to each knee were evaluated three times at upright kneeling (UK) and full kneeling (FK) positions, in different ankle conditions (dorsiflexion and plantarflexion) with static balance device. HurSmart balance system (HUR smart balance, HUR, Helsinki, Finland) was used for assessed the weight distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No